CLINICAL TRIAL: NCT05393570
Title: Partnering Lifestyle Intervention With Bariatric Surgery to Maximize Health Outcomes in Adolescents
Brief Title: Lifestyle Improvement for Teens With Bariatric Surgery
Acronym: LIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sarah E Messiah, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-SPH-19-0406; 1R21HD105129-01A1 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2022-05-26 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Obesity, Adolescent; Bariatric Surgery Candidate
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Behavioral: Healthy Lifestyle Behavioral Intervention (MBS -supported intervention)

INTERVENTIONS:
Behavioral: Healthy Lifestyle Behavioral Intervention (MBS -supported intervention) — After patient/parent consent is completed, participants will begin the pre-MBS intervention phase. A minimum of 6 1- hour sessions will occur pre-MBS, and 26 will occur post-MBS.Dr. Klement, MBS coordinator and a diabetes educator will manage session delivery to adolescents/parents. All content will follow the Diabetes Prevention Program (DPP)-adapted curriculum flow. After that the research assistant will perform outreach, reminder calls, and follow-up for missed appointments. Pre-and post-MBS intervention delivery (based on adapted curriculum/model) may consist of a combination of 1-on-1 and group sessions (in-person or virtually), and online support tools, dependent upon adolescent/parent qualitative feedback on delivery method preference.

SUMMARY:
This study aims to conduct a proof-of-concept study to assess the feasibility, acceptability, and effectiveness of a Metabolic and bariatric surgery (MBS) -supported healthy lifestyle behavioral intervention among adolescent patients, their families, and their clinical team.

DETAILED DESCRIPTION:
This proof-of-concept study aims to evaluate the feasibility, acceptability, and preliminary effectiveness of a lifestyle behavioral intervention integrated with metabolic and bariatric surgery (MBS) for adolescents with severe obesity. Targeting youth aged 12-18, the intervention is designed to enhance pre- and post-operative outcomes by supporting sustained healthy behaviors among patients and their families. Guided by formative qualitative research (AIM 1), the team will adapt an evidence-based multimedia lifestyle program (AIM 2) to align with adolescent MBS patients' unique needs and preferences.

The adapted intervention will then be pilot-tested (AIM 3) among adolescent patients at a large adolescent healthcare system, with participants followed up to 12 months post-surgery. The program includes online components delivered before and after surgery, with progress evaluated at multiple time points. In addition to anthropometric and cardiometabolic outcomes, the study will assess intervention engagement, satisfaction, and delivery fidelity using the RE-AIM framework. The overarching goal is to demonstrate that combining lifestyle support with MBS can improve adherence, reduce attrition, and enhance long-term health outcomes among adolescents with severe obesity.

ELIGIBILITY:
Inclusion Criteria

* Must meet National Institutes of Health criteria to qualify for MBS for adolescents (BMI >35 kg/m^2 and at least one existing co-morbidity [e.g. elevated blood pressure, hypercholesterolemia, etc.] or a BMI>40kg/m^2).
* received psychological clearance for surgery

Exclusion Criteria:

* is not medically referred by a physician for bariatric surgery
* Refuses to participate in the study

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Messiah, Ph.D., MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescents were recruited from a single tertiary care center MBS program. Additionally, the clinic staff provided MBS program patient lists in EPIC. Adolescents were eligible if they met the National Institute of Health criteria for MBS, could communicate in English or Spanish, were between 12 and 18 years old, and had stable internet access or could access materials via smartphones. All participants underwent Laparoscopic Sleeve Gastrectomy.
Groups:
- Treatment: Adolescents who met the inclusion/exclusion criteria and consented to be participants in the study.
  Inclusion Criteria
  Must meet National Institutes of Health criteria to qualify for MBS for adolescents (BMI >35 kg/m2 and at least one existing co-morbidity [e.g., elevated blood pressure, hypercholesterolemia, etc.] or a BMI>40kg/m2).
  Received psychological clearance for surgery
  Exclusion Criteria:
  Is not medically referred by a physician for bariatric surgery Refuses to participate in the study
Period: Overall Study
Arm/Group | Treatment
Started | 76
Completed | 29
Not Completed | 47

BASELINE CHARACTERISTICS:
Population: Adolescents who met the inclusion/exclusion criteria and consented to be participants in the study.
  Inclusion Criteria
  Must meet National Institutes of Health criteria to qualify for MBS for adolescents (BMI >35 kg/m2 and at least one existing co-morbidity [e.g., elevated blood pressure, hypercholesterolemia, etc.] or a BMI>40kg/m2).
  Received psychological clearance for surgery
  Exclusion Criteria:
  Is not medically referred by a physician for bariatric surgery Refuses to participate
Groups:
- Treatment: Adolescents who met the inclusion/exclusion criteria and consented to be participants in the study.
  Inclusion Criteria
  Must meet National Institutes of Health criteria to qualify for MBS for adolescents (BMI >35 kg/m^2 and at least one existing co-morbidity [e.g., elevated blood pressure, hypercholesterolemia, etc.] or a BMI>40kg/m^2).
  Received psychological clearance for surgery
  Exclusion Criteria:
  Is not medically referred by a physician for bariatric surgery Refuses to participate in the study
Arm/Group | Treatment
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants] — Years (Self-reported)
  Participants
    <=18 years | 76
    Between 18 and 65 years | 0
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] — Years (Self-reported)
  Years | 15.67 (1.37)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex (Self-reported)
  Participants
    Female | 53
    Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity (Self-reported)
  Participants
    Hispanic or Latino | 43
    Not Hispanic or Latino | 29
    Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race (Self-reported)
  Participants
    American Indian or Alaska Native | 1
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 1
    Black or African American | 23
    White | 27
    More than one race | 24
    Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI (kg/m2) at enrollment
  kg/m^2 | 48.27 (8.32)

OUTCOME MEASURES:

1. Primary Outcome: Change in Health-related Quality of Life as Measured by the HRQOL-14
Description: This survey includes 3 modules (Healthy Days Core Module = 4 questions, Activity Limitations Module = 5 questions, and the Healthy Days Symptoms Module = 5 questions). This survey is not based on a summary score. Instead to evaluate the score unhealthy days are the estimated total number of days in a 30 day period where participants felt their physical or mental health was not good. Survey responses from question 2 and 3 in the Healthy Days Core Module are combined to get overall unhealthy days.
Time Frame: Pre-surgery, 6 months post-surgery
Measure: Mean (Standard Deviation); unit: days
Groups:
- MBS Completers: Adolescents who met the inclusion/exclusion criteria, consented to be participants in the study, and received MBS while participating in the study.
Arm/Group | MBS Completers
Number analyzed (Participants) | 29
days | -9 (19.04)

2. Primary Outcome: Change in Blood Lipid Levels as Assessed by Lipid Panel
Description: Cholesterol (mg/dL), HDL cholesterol (mg/dL), Triglycerides (mg/dL), LDL cholesterol (mg/dL), non-HDL cholesterol (mg/dL) change from pre-surgery to 6 months post-surgery.
Time Frame: Pre surgery, 6 months post surgery
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MBS Completers
Number analyzed (Participants) | 29
mg/dL
  Cholesterol | -3.97 (23.22)
  HDL cholesterol | 4.36 (7.55)
  Triglycerides | -45.36 (42.70)
  LDL cholesterol | 0.82 (16.07)
  non-HDL cholesterol | -8.18 (21.93)

3. Primary Outcome: Change in Blood Glucose Level
Description: Measure of Blood Glucose (mg/dL) change from pre-surgery to 6 months post-surgery.
Time Frame: pre surgery, 6 months post surgery
Measure: Mean (Standard Deviation); unit: (mg/dL)
Arm/Group | MBS Completers
Number analyzed (Participants) | 29
(mg/dL) | -2.3 (11.17)

4. Primary Outcome: Change in Diastolic Blood Pressure
Description: Measure diastolic blood pressure (mmHg) change from pre-surgery to 6 months post-surgery.
Time Frame: pre surgery, 6 months post surgery
Measure: Mean (Standard Deviation); unit: (mmHg)
Arm/Group | MBS Completers
Number analyzed (Participants) | 29
(mmHg) | -5 (12.50)

5. Primary Outcome: Change in Systolic Blood Pressure
Description: Measure systolic blood pressure (mmHg) change from pre-surgery to 6 months post-surgery.
Time Frame: pre surgery, 6 months post surgery
Measure: Mean (Standard Deviation); unit: (mmHg)
Arm/Group | MBS Completers
Number analyzed (Participants) | 29
(mmHg) | -3.81 (16.22)

6. Primary Outcome: Change in HbA1c Levels
Description: Measure HbA1c% (mmol/mol) levels in blood change from pre-surgery to 6 months post-surgery.
Time Frame: pre surgery, 6 months post surgery
Measure: Mean (Standard Deviation); unit: (mmol/mol)
Arm/Group | MBS Completers
Number analyzed (Participants) | 29
(mmol/mol) | -0.353 (0.297)

ADVERSE EVENTS:
Time Frame: Enrollment to 6-month post-surgery
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76
Other Adverse Events (participants affected / at risk) | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT05393570/Prot_SAP_000.pdf